CLINICAL TRIAL: NCT06361498
Title: Accuracy of Ultrasound for the Evaluation of Percutaneous Gastrostomy Tube Position and Leakage
Brief Title: Ultrasound for Evaluation of Percutaneous G-tube Position
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 23-3115
Record Dates: First submitted 2024-03-22; First posted 2024-04-12 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Gastrostomy
Keywords: gastrostomy tube; ultrasound; fluoroscopy
MeSH Terms: interventions — Ultrasonography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Ultrasound Imaging (Other): This study consists of one group/ All participants will receive ultrasound imaging prior to the standard of care fluoroscopic imaging.
  Interventions: Device: Ultrasound Imaging

INTERVENTIONS:
Device: Ultrasound Imaging — Participant will receive ultrasound imaging to evaluate the replaced G-tube placement.

SUMMARY:
The goal of this clinical trial is to compare using ultrasound imaging to look at the position of the gastrostomy tube (GT) against fluoroscopic imaging in pediatric patients who had a recent GT tube replacement.

The main questions it aims to answer are:

* If ultrasound is just as accurate as fluoroscopy to assess the GT position.
* If ultrasound takes less time than fluoroscopy to assessing the GT position.

Participants will be imaging using ultrasound to assess GT positioning before their standard of care fluoroscopic imaging.

DETAILED DESCRIPTION:
This clinical trial will address the validity of using ultrasound to evaluate the position of the gastrostomy tube (GT) retention balloon against the clinical gold standard of fluoroscopic tube injection to assess for potential larger studies and the implementation in clinical practice. This study will address the ability to visualize the retention balloon within the gastric lumen, the ability to assess for leakage from the GT within the abdomen, and the relative length of each study to perform.

ELIGIBILITY:
Inclusion Criteria:

An individual who presents with a dislodged GT and meets one of the following minor criteria:

* Surgical GT placement less than 90 days from presentation
* Traumatic GT dislodgement/removal
* Recent stoma dilation
* Clinician uncertainty about position of GT placement

Exclusion Criteria:

* An individual >18 years of age
* Acutely ill patients defined as hemodynamically unstable defined as any child who has abnormal vital signs or disruption of vital functions (i.e. airway, breathing, circulation, mental function). Vital signs are based on patient age. Initial assessment of clinical patient stability will be provided by the ordering/referring provider.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-04-30 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Proportion of Ultrasound that Agree with Fluoroscopy with Respect to Identifying the GT Location | Upon completion of all study image data collection for all participants [approximately 1 year]
  Proportional accuracy of ultrasound in identifying the gastrostomy tube (GT) balloon location based on the readers' (radiologists) ability to use the ultrasound to locate the GT balloon in comparison with the gold standard (fluoroscopic tube injection).

SECONDARY OUTCOMES:
Sensitivity of ultrasound (US) to determine the visualization of GT leakage | Upon completion of all study image data collection for all participants [approximately 1 year]
  Sensitivity of ultrasound to determine the visualization of the GT leakage is defined as the ability of readers (radiologists) to use the ultrasound to determine the presence or absence of injected saline leakage under ultrasound using fluoroscopic tube injection as the gold standard.
Specificity of ultrasound (US) to determine the visualization of GT leakage | Upon completion of all study image data collection for all participants [approximately 1 year]
  Specificity of ultrasound to determine the visualization of the GT leakage is defined as the ability of readers (radiologists) to use the ultrasound to determine the presence or absence of injected saline leakage under ultrasound using fluoroscopic tube injection as the gold standard.
Duration of ultrasound (US) to complete evaluation of GT position | Upon completion of all study image data collection for all participants [approximately 1 year]
  Duration of ultrasound to complete the evaluation of the GT position is defined as the length of time necessary to complete a research US evaluation of the GT position using fluoroscopic tube injection as the gold standard.

CONTACTS AND LOCATIONS:
Overall Officials: William Pryor, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.
Supporting Information: Study Protocol
Time Frame: 9 to 36 months following publication.
Access Criteria: The investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.